CLINICAL TRIAL: NCT05899387
Title: Prospective, International, Multicenter Minimal Interventional Study to Detect Possible Markers for Prediction of Seroma Development and Risk Assessment of a Breast Seroma After Mastectomy with or Without Implant-based Breast Reconstruction
Brief Title: Seroma of the Mammary Gland
Acronym: SerMa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Principal Investigator, Nina Ditsch, Prof. Dr. med., University Hospital Augsburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1.0
Record Dates: First submitted 2023-02-07; First posted 2023-06-12 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Seroma; Breast Cancer; Mastectomy; Breast Implant; Complications
MeSH Terms: conditions — Seroma; Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- BC, mastectomy and implant (Experimental): Women with first diagnosis of breast cancer or DCIS and planned skin-sparing mastectomy and implant placement
  Interventions: Procedure: Swap collection; Procedure: Seroma punction; Procedure: Blood sampling; Diagnostic Test: Sonographic correlation Seroma
- BC and mastectomy (Active Comparator): Women with first diagnosis of breast cancer or DCIS and planned simple mastectomy
  Interventions: Procedure: Swap collection; Procedure: Seroma punction; Procedure: Blood sampling; Diagnostic Test: Sonographic correlation Seroma
- High risk for BC (Active Comparator): healthy women with high risk for breast cancer and planned bilateral risk-reducing mastectomy and implant reconstruction
  Interventions: Procedure: Swap collection; Procedure: Seroma punction; Procedure: Blood sampling; Diagnostic Test: Sonographic correlation Seroma
- Cosmetic breast surgery (Active Comparator): healthy women planned for plastic breast implant surgery
  Interventions: Procedure: Swap collection; Procedure: Seroma punction; Procedure: Blood sampling; Diagnostic Test: Sonographic correlation Seroma

INTERVENTIONS:
Procedure: Swap collection — Performing the surgery (Mastectomy with or without implant reconstruction; Insertion of Breast implants for control group 3) according to valid standards.
  In addition, taking swabs intraoperatively according to protocol from skin and surgical site.
Procedure: Seroma punction — Puncturing of a seroma in case of occurence and clinical need
Procedure: Blood sampling — Blood sampling at defined time points according to protocol
Diagnostic Test: Sonographic correlation Seroma — If a seroma occurs, a sonographic correlation is performed to determine the exact size of the seroma

SUMMARY:
The study is designed as international, prospective, minimal interventional study in cooperation with EUBREAST e.V. (European Breast Cancer Research Association of Surgical Trialists). Furthermore, it is planned to initiate a registry for postoperative breast seromas.

DETAILED DESCRIPTION:
Postoperative seroma formations are one of the most common and serious complications after breast surgery, above all after mastectomy. Especially in patients who have opted for breast reconstruction using implants, seromas lead to infections and wound dehiscence which can result in implant and finally breast loss. To date, the cause of seroma development has not yet been clarified. First data of a pilot study of our research group identified an association with immunological-inflammatory processes as a possible cause for seroma development (Seroma after Simple Mastectomy in Breast Cancer-The Role of CD4+ T Helper Cells and the Evidence as a Possible Specific Immune Process; Pochert et al. 2022).

The main objective of the SerMa (Seroma of the Mammary gland) study presented here is to identify patient groups who have an increased risk of developing seromas based on immunological/inflammatory processes. Based on the findings clinical consequences should be developed in the future, such as more precise risk-adapted patient education and individualized advising regarding the selection of the reconstruction procedure, with the goal of minimizing complication rates. In addition, analyses of the tumor and the microenvironment will be performed to differentiate possible carcinoma-specific immunological processes.

ELIGIBILITY:
Inclusion criteria study group and control group 1:

* Written informed consent
* Age ≥ 18 years
* all stages of DCIS or primary breast cancer (T1-T4, N0 or N+, M0) including all histopathological subtypes (ER/PR positive, ER positive/PR negative, Her-2/neu positive and triple negative)
* Surgical procedure planned including ablatio or subcutaneous mastectomy with implant or expander insertion

Inclusion criteria control group 2 and 3:

* Written informed consent
* Age ≥ 18 years
* Surgical procedure planned with implant or expander insertion with or without subcutaneous mastectomy

Exclusion criteria:

* Age <18 years
* Male sex
* Breast cancer patients planned for breast conserving therapy
* Recurrent breast cancer disease
* History of breast surgery
* Diagnosis of LCIS only
* Pregnancy at time of diagnosis
* Patients with a known immunodeficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Identification of a patient population at increased risk for developing seroma. | Follow-up for each participant: 6 month
  * Examination of seroma fluid and blood samples to identify immunological markers.
  * Local microbiome analyses to investigate a possible bacterial colonization.
  * Tissue analyses to determine possible carcinoma-specific immunologic processes.

SECONDARY OUTCOMES:
Comparison of findings in local and systemic measurements in patients with and without seroma. | Follow-up for each participant: 6 month
Comparison of the groups with or without cancer regarding development of seroma. | Follow-up for each participant: 6 month
Comparison of the clinicopathologic differences between the implant and simple mastectomy group within both cancer groups | Follow-up for each participant: 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Kühn, Prof., Study Chair — Eubreast Network, Baumreute 37 D-73730 Esslingen, Germany; Nina Ditsch, Prof., Principal Investigator — University Hospital Augsburg, Stenglinstr. 2, D-86156 Augsburg, Germany
Locations (1):
- University Hospital Augsburg, Department of Gynecology and Obstetrics, Augsburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No